CLINICAL TRIAL: NCT06530641
Title: Evaluation of Clinical Impact of the Type of Cardioplegia Used in the Patient Undergoing Major Cardiac Surgery with Extracorporeal Circulation. CARDIO-HEART Clinical Trial.
Brief Title: Evaluation of Clinical Impact of the Type of Cardioplegia Used in the Patient Undergoing Major Cardiac Surgery.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lourdes Montero Cruces (Other)
Responsible Party: Sponsor-Investigator, Lourdes Montero Cruces, Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24/238-EC_M
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Surgery; Cardioplegia; Heart Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Once the patient is included in the study, they will be assigned an identification number and a treatment group.
  * Group 1: Patients who will be administered Buckberg blood cardioplegia.
  * Group 2: Patients who will be administered Custodiol crystalloid cardioplegia. A 1:1 randomization will be carried out by blocks and stratified by weight of the intervention according to the EuroSCORE II:
    * Weight 1: Any major cardiac procedure (40% of the sample).
    * Weight 2: Two major cardiac procedures (40% of the sample).
    * Weight 3: Three or more major cardiac procedures (20% of the sample).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buckberg (Active Comparator): Patients who will be administered Buckberg blood cardioplegia.
  Interventions: Drug: Buckberg Cardi-Braun
- Custodiol (Experimental): Patients who will be administered Custodiol crystalloid cardioplegia.
  Interventions: Drug: Custodiol Htk Soln

INTERVENTIONS:
Drug: Custodiol Htk Soln — Patients undergoing major cardiac surgery with extracorporeal circulation who are administered Custodiol crystalloid cardioplegia.
  Other Names: Custodiol HTK solution. ACT: K944866
  Arms: Custodiol
Drug: Buckberg Cardi-Braun — Patients undergoing major cardiac surgery with extracorporeal circulation who are administered Buckberg blood cardioplegia.
  Other Names: Buckberg Cardi-Braun cardioplegia solution. ATC: B05X A16.
  Arms: Buckberg

SUMMARY:
Phase IV clinical trial of a single-blind, prospective and longitudinal randomized intervention comparing patients undergoing major cardiac surgery with extracorporeal circulation who are administered Custodiol crystalloid cardioplegia versus Buckberg blood cardioplegia.

DETAILED DESCRIPTION:
Myocardial protection by administering cardioplegia is a fundamental concept during cardiopulmonary bypass in patients undergoing cardiac surgery. It is a multifactorial strategy, in which cardioplegia is the most important. To date, there is no standardized consensus on the use of cardioplegia in different cardiac surgery procedures, and the best strategy continues to be debated given the wide range available. The choice of the type of cardioplegia should be made on an individual basis, taking into account the surgical procedure and clinical context. The need for a single dose of cardioplegia could favor the use of Custodiol crystaloid cardioplegia in complex cardiac surgeries that require longer extracorporeal circulation time. Both cardioplegia are safe and effective and widely used globally; however, the information provided in the literature is limited, with most of the information coming from retrospective studies.The objective of the present study is to demonstrate the non-inferiority of Custodiol crystalloid cardioplegia versus Buckberg blood cardioplegia in patients undergoing major cardiac surgery with extracorporeal circulation with prolonged aortic clamping times.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with cardiac pathology and indication for major cardiac surgery with extracorporeal circulation and aortic clamping.

Exclusion Criteria:

1. Pregnancy.
2. Aortic arch procedures.
3. Procedures in which hypothermia <28ºC is expected during the intervention.
4. Minimally invasive procedures "Port Access".
5. Active endocarditis.
6. Emerging procedures.
7. Isolated aortic valve replacements.
8. Decision of the main surgeon not to participate in the study due to other clinical criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the composite event | 90 days after the intervention
  Comparison of the composite event of death, perioperative AMI, low cardiac postoperative output with need for ionotropics, and AKIN-III acute kidney failure

SECONDARY OUTCOMES:
Differences in the incidence of elevation of Troponin | 90 days after the intervention
  Comparison of the elevation of Troponin I US at 12 and 24 hours after the procedure.
Differences in the 90-day mortality rate | 90 days after the intervention
  Comparison of 90-day postoperative mortality
Differences in the incidence of low cardiac postoperative output | 90 days after the intervention
  Comparison of low cardiac postoperative output event with need for ionotropic drugs in the first 24 hours.
Differences in the incidence of acute kidney failure event | 90 days after the intervention
  Comparison of AKIN-III acute kidney failure event
Differences in the incidence of acute myocardial infarction | 90 days after the intervention
  Comparison of perioperative AMI incidence
Differences in the incidence of major bleeding event | 90 days after the intervention
  Comparison of major bleeding event or life-threatening or disabling hemorrhage.
Differences in the incidence of the need of transfusion | 90 days after the intervention
  Comparison of the need for transfusion of blood products (absolute number) in the first 48 hours.
Differences in the incidence of prolonged mechanical ventilation | 90 days after the intervention
  Comparison of the need for prolonged mechanical ventilation for >24h.
Differences in the incidence of neurological complications | 90 days after the intervention
  Comparison of type 1 and type 2 neurological complications.
Differences in the incidence of postoperative atrial fibrillation. | 90 days after the intervention
  Comparison of the incidence of postoperative atrial fibrillation.
Differences in the overall survival rate at 90 days. | 90 days after the intervention
  Comparison of overall survival at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Montero Cruces, Principal Investigator — Hospital San Carlos, Madrid
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No